CLINICAL TRIAL: NCT04355221
Title: Pulsed Radiofrequency in Treatment of Classic Trigeminal Neuralgia (Prolonged Duration Versus Higher Voltage)
Brief Title: Pulsed Radiofrequency in Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD/16.06.26
Record Dates: First submitted 2019-12-01; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Trigeminal Neuralgia
Keywords: pulsed radiofrequency
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): using the standard settings of pulsed radiofrequency technique (PRFT). two cycles, each one for 2 minutes at 45 Volts (V) with a pulse width of 10 milliseconds (ms) and a pulse frequency of 4 Hertz (Hz). The cut-off needle tip temperature is set at 420 Celsius (C).
  Interventions: Procedure: pulsed radiofrequency
- Group B (Experimental): using prolonged duration of PRFT. four cycles, each one for 2 minutes at 45V with a pulse width of 10ms and a pulse frequency of 4Hz. The cut-off needle tip temperature is set at 420C.
  Interventions: Procedure: pulsed radiofrequency
- Group C (Experimental): using higher voltage PRFT.. two cycles, each one for 2 minutes at 60V with a pulse width of 10ms and a pulse frequency of 4Hz. The cut-off needle tip temperature is set at 420C.
  Interventions: Procedure: pulsed radiofrequency

INTERVENTIONS:
Procedure: pulsed radiofrequency — Pulsed radiofrequency of the trigeminal nerve using NeuroTherm NT 1100 RF generator device

SUMMARY:
The current study investigated the efficacy of pulsed radiofrequency in pain reduction in TN patients and compared the efficacy and the impact on the quality of life of the standard technique with a prolonged duration technique and a higher voltage one.

Entire enrolled patients were diagnosed as classic TN according to the international headache society classification (IHS, 2013) and underwent brain MRI and MRA to exclude secondary causes. Patients were randomly divided into three groups, Group A patients underwent PRF using the standard settings, group B patients underwent PRF with prolonged duration and Group C patients underwent PRF with higher voltage. VAS and pain amplitude reduction were recorded before the intervention and 1 hour, 1 day, 1week, 1 month, 6 months and 1year after it. Quality of life was assessed before and 1 year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed as classic TN according to the international headache society classification of headache disorders
* Visual analogue scale (VAS) for pain of at least 4 or more.
* Pain is refractory to medical treatment (for at least 3 months with three drugs including carbamazepine with optimum dosage) or patients who developed intolerable side effects from medications.

Exclusion Criteria:

* Symptomatic (secondary) TN: which is causes by structural lesion other than neurovascular compression such as multiple sclerosis, tumors, stroke or trauma according to the international headache society classification (IHS, 2013).

Local infection at the site of the needle puncture. Bleeding tendency or coagulopathy. Previous treatment with invasive treatments such as radiofrequency thermo coagulation, destructive chemical injection, gamma knife treatment, percutaneous balloon micro-compression or microvascular decompression.

Major mental or psychiatric disorders. History of drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Pain amplitude reduction | 1 year
  compare the pain amplitude reduction in the three groups using the visual analogue pain scale

SECONDARY OUTCOMES:
RAND 36-Item Health Survey | 1 year
  compare the quality of life changes before and after intervention using RAND 36-Item Health Survey

IPD SHARING:
Plan to Share IPD: Undecided